CLINICAL TRIAL: NCT04362137
Title: Phase 3 Randomized, Double-blind, Placebo-controlled Multi-center Study to Assess the Efficacy and Safety of Ruxolitinib in Patients With COVID-19 Associated Cytokine Storm (RUXCOVID)
Brief Title: Study to Assess the Efficacy and Safety of Ruxolitinib in Patients With COVID-19 Associated Cytokine Storm
Acronym: RUXCOVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CINC424J12301; INCB 18424-368 (Other: Incyte Study Code); 2020-001662-11 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Cytokine Storm (Covid-19)
Keywords: COVID-19 pneumonia; cytokine release syndrome; SARS-COV-2; ruxolitinib
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib 5 mg (Experimental): Ruxolitinib 5 mg tablets twice daily (b.i.d.) for 14 days with possible extension of treatment to 28 days
  Interventions: Drug: Ruxolitinib
- Placebo (Placebo Comparator): Matching-image placebo for 14 days with possible extension of treatment to 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 5 mg tablets
  Other Names: INC424
  Arms: Ruxolitinib 5 mg
Drug: Placebo — Matching-image placebo
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled, 29-day, multicenter study to assess the efficacy and safety of ruxolitinib + standard-of-care (SoC) therapy, compared with placebo + SoC therapy, in patients aged ≥12 years with COVID-19 disease.

DETAILED DESCRIPTION:
This was a Phase III, multicenter, double-blind, randomized, placebo-controlled study to assess the efficacy and safety of ruxolitinib in patients aged ≥12 years with COVID-19 disease. The study enrolled patients to ruxolitinib or placebo, in addition to standard of care (SoC) per local practice. Patients who meet the inclusion/exclusion criteria were randomized in a 2:1 ratio to either oral ruxolitinib 5 mg twice daily + SoC or oral matching-image placebo + SoC for a total of 14 days. An additional 14 days of study drug could be given if in the opinion of the investigator the patient's clinical signs and symptoms did not improve, or worsen, and the potential benefit outweighed the potential risk.

The study included:

* Screening period of 0-2 days.
* Study period of 29 days (treatment of 14 days with possible extension of treatment to 28 days).

The primary objective was to evaluate the efficacy (as measured by a composite endpoint of proportion of patients who die, develop respiratory failure [require mechanical ventilation], or require intensive care unit care) of ruxolitinib + standard-of-care (SoC) therapy compared with placebo + SoC therapy, for the treatment of COVID-19 by Day 29.

ELIGIBILITY:
Inclusion Criteria:

Patient or guardian/health proxy must provide informed consent (and assent if applicable) before any study assessment is performed.

Male and female patients aged ≥ 12 years (or ≥ the lower age limit allowed by Health Authority and/or Ethics Committee/Institutional Review Board approvals).

Patients with coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) test or another rapid test from the respiratory tract prior to randomization.

Patients currently hospitalized or will be hospitalized prior to randomization.

Patients, who meet at least one of the below criteria:

* Pulmonary infiltrates (chest X ray or chest CT scan);
* Respiratory frequency ≥ 30/min;
* Requiring supplemental oxygen;
* Oxygen saturation ≤ 94% on room air;
* Arterial oxygen partial pressure (PaO2)/ fraction of inspired oxygen (FiO2) < 300mmHg (1mmHg=0.133kPa) (corrective formulation should be used for higher altitude regions (over 1000m).

Exclusion Criteria:

History of hypersensitivity to any drugs or metabolites of similar chemical classes as ruxolitinib.

Presence of severely impaired renal function defined by serum creatinine > 2 mg/dL (>176.8 μmol/L), or have estimated creatinine clearance < 30 ml/min measured or calculated by Cockroft Gault equation or calculated by the updated bedside Schwartz equation.

Suspected uncontrolled bacterial, fungal, viral, or other infection (besides COVID-19).

Currently intubated or intubated between screening and randomization. In intensive care unit (ICU) at time of randomization. Intubated or in ICU for COVID-19 disease prior to screening. Patients who are on anti-rejection, immunosuppressant or immunomodulatory drugs (i.e. tocilizumab, ruxolitinib, canakinumab, sarilumab, anakinra).

Unable to ingest tablets at randomization. Pregnant or nursing (lactating) women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (11):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Idaho Falls, Idaho
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, C A B A, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Brazil (5):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Colombia (3):
  - Novartis Investigative Site, Rionegro, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
- France (5):
  - Novartis Investigative Site, Colombes
  - Novartis Investigative Site, Eaubonne
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Pierre-Bénite
- Germany (3):
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
- Mexico (3):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Mexico City, Mexico CP
  - Novartis Investigative Site, Estado de México
- Peru (3):
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Lima
- Russia (6):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
- Spain (4):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (4):
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Han MK, Antila M, Ficker JH, Gordeev I, Guerreros A, Bernus AL, Roquilly A, Sifuentes-Osornio J, Tabak F, Teijeiro R, Bandelli L, Bonagura DS, Shu X, Felser JM, Knorr B, Cao W, Langmuir P, Lehmann T, Levine M, Savic S. Ruxolitinib in addition to standard of care for the treatment of patients admitted to hospital with COVID-19 (RUXCOVID): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Rheumatol. 2022 May;4(5):e351-e361. doi: 10.1016/S2665-9913(22)00044-3. Epub 2022 Mar 29. PMID 35368384
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 61 investigative sites in 12 countries.
Pre-assignment Details: Patients were to be randomized on the same day as screening or up to 2 days after completing the screening procedures.
Period: Overall Study
Arm/Group | Ruxolitinib 5 mg | Placebo
Started (Randomized participants.) | 287 | 145
Safety Set (The Safety Set included all participants who received at least one dose of double-blind treatment.) | 281 | 143
Completed | 269 | 139
Not Completed | 18 | 6
Not completed — Death | 9 | 3
Not completed — Patient decision | 6 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib 5 mg | Placebo | Total
Number analyzed (Participants) | 287 | 145 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (13.7) | 56.9 (12.5) | 56.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 72 | 197
  Male | 162 | 73 | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 242 | 109 | 351
  American Indian Or Alaska Native | 26 | 13 | 39
  Black Or African American | 6 | 9 | 15
  Asian | 5 | 5 | 10
  Multiple | 3 | 2 | 5
  Unknown | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Die, Develop Respiratory Failure [Require Mechanical Ventilation] or Require Intensive Care Unit (ICU) Care
Description: Efficacy is measured by a composite endpoint of proportion of patients who die, develop respiratory failure [require mechanical ventilation], or require intensive care unit [ICU] care for the treatment of COVID-19. Analyses are cumulative, thus analysis on Day 29 includes all events till that day. Patients who developed respiratory failure and/or required ICU at randomization are excluded from the analysis.
Time Frame: Day 1 - Day 29
Population: Randomized participants excluding those who developed respiratory failure and/or required ICU at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 284 | 144
Participants | 34 | 17
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Test type: Superiority; p = 0.769, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.48 to 1.73] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm

2. Secondary Outcome: Clinical Status
Description: Clinical status is measured with the 9-point ordinal scale.
  The scoring is:
  * Uninfected patients have a score 0 (no clinical or virological evidence of infection).
  * Ambulatory patients (not in hospital or in hospital and ready for discharge) can have a score 1 (no limitation of activities) or 2 (limitation of activities).
  * Hospitalized patients with mild disease can have score 3 (no oxygen therapy defined as peripheral oxygen saturation (SpO2) ≥ 94% on room air) or 4 (oxygen by mask or nasal prongs).
  * Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)).
  * Patients who die have a score 8.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
score on scale
  Baseline: number analyzed (Participants) | 286 | 145
  Baseline | 3.7 (0.56) | 3.7 (0.53)
  Day 15: number analyzed (Participants) | 280 | 142
  Day 15 | 1.8 (1.54) | 1.8 (1.41)
  Day 29: number analyzed (Participants) | 278 | 142
  Day 29 | 1.1 (1.61) | 1.0 (1.41)

3. Secondary Outcome: Percentage of Patients With at Least Two-point Improvement From Baseline in Clinical Status
Description: Percentage of patients with at least two points improvement in clinical status on the 9-point ordinal scale. The baseline value of clinical status is defined as the last assessment prior to first dose of double-blind treatment. Patients with missing data at Day 15 and/or Day 29 are treated as non-responders.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment of clinical status at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
Participants
  Day 15 | 206 | 108
  Day 29 | 252 | 129
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.647, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.55 to 1.46] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; p = 0.997, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.52 to 1.92] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm

4. Secondary Outcome: Percentage of Patients With at Least One-point Improvement From Baseline in Clinical Status
Description: Percentage of patients with at least one point improvement in clinical status on the 9-point ordinal scale. The baseline value of clinical status is defined as the last assessment prior to first dose of double-blind treatment. Patients with missing data at Day 15 and/or Day 29 are treated as non-responders.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment of clinical status at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
Participants
  Day 15 | 250 | 128
  Day 29 | 261 | 136
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.946, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.51 to 1.87] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; p = 0.573, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.35 to 1.79] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm

5. Secondary Outcome: Percentage of Patients With at Least One-point Deterioration From Baseline in Clinical Status
Description: Percentage of patients with at least one point deterioration in clinical status on the 9-point ordinal scale. The baseline value of clinical status is defined as the last assessment prior to first dose of double-blind treatment. Patients with missing data at Day 15 and/or Day 29 are treated as non-responders.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment of clinical status at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
Participants
  Day 15 | 16 | 9
  Day 29 | 14 | 5
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.532, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.31 to 1.83] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; p = 0.764, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.40 to 3.49] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm

6. Secondary Outcome: Time to Improvement in Clinical Status
Description: Time to improvement in clinical status from baseline category to one less severe category of the 9-point ordinal scale. The baseline value of clinical status is defined as the last assessment prior to first dose of double-blind treatment.
  Median time to improvement is estimated by Kaplan-Meier method, with dead patients being censored at the maximum follow-up time in the study. Patients who did not achieve improvement and did not die are censored at their last clinical status assessment date.
Time Frame: 29 days
Population: Randomized participants with a valid assessment of clinical status at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
days | 9.0 [8.0 to 10.0] | 9.0 [8.0 to 12.0]
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Test type: Superiority; p = 0.330, Proportional hazards model; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.90 to 1.37] — Between group comparison using competing risk framework. A hazard ratio > 1 favors the ruxolitinib 5 mg arm

7. Secondary Outcome: Mean Change From Baseline in the Clinical Status
Description: Mean change from baseline in the 9-point ordinal scale. The baseline value of clinical status is defined as the last assessment prior to first dose of double-blind treatment. Patients with missing data at Day 15 and/or Day 29 are excluded from the analysis.
  A negative change from baseline in the clinical status is a favorable outcome.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
score on scale
  Day 15: number analyzed (Participants) | 280 | 142
  Day 15 | -1.96 (0.084) | -1.93 (0.118)
  Day 29: number analyzed (Participants) | 278 | 142
  Day 29 | -2.61 (0.090) | -2.69 (0.126)
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.831, ANCOVA; Least squares (LS) mean = -0.03, 95% CI 2-sided [-0.31 to 0.25], Standard Error of Mean 0.144
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; p = 0.624, ANCOVA; LS Mean = 0.08, 95% CI 2-sided [-0.23 to 0.38], Standard Error of Mean 0.155

8. Secondary Outcome: Mortality Rate
Description: Mortality rate is determined as the proportion of participants who died by study Day 15 and Day 29
Time Frame: Day 15, Day 29
Population: All randomized participants including those who did not receive any dose, as per intent-to-treat principle, and excluding patients lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
Participants
  Day 15: number analyzed (Participants) | 286 | 145
  Day 15 | 6 | 2
  Day 29: number analyzed (Participants) | 286 | 145
  Day 29 | 9 | 3
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.944, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.20 to 5.57] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; p = 0.775, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.35 to 5.11] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm

9. Secondary Outcome: Proportion of Patients Requiring Mechanical Ventilation
Description: Proportion of patients requiring mechanical ventilation. Analyses are cumulative, thus analysis on Day 29 includes all events till that day. Patients who required mechanical ventilation at randomization are excluded from the analysis.
Time Frame: Day 1 - Day 29
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
Participants | 22 | 10
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Test type: Superiority; p = 0.987, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.45 to 2.21] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio < 1 favors the ruxolitinib 5 mg arm

10. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization is defined as time to hospital discharge. Median time to hospital discharge is estimated by Kaplan-Meier method, with dead patients being censored at the maximum follow-up time in the study. Patients who were not discharged and did not die are censored at their last assessment date.
Time Frame: 29 days
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
days | 9.0 [8.0 to 10.0] | 9.0 [8.0 to 12.0]
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Test type: Superiority; p = 0.738, Proportional hazards model; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.84 to 1.28] — Between group comparison using competing risk framework. A hazard ratio > 1 favors the ruxolitinib 5 mg arm

11. Secondary Outcome: Time to Hospital Discharge or to a NEWS2 Score of ≤2
Description: The time to hospital discharge or to a National Early Warning Score 2 (NEWS2) of ≤2 and maintained for 24 hours whichever comes first.
  The NEWS2 is based on a simple aggregate scoring system in which a score is allocated to physiological measurements, already recorded in routine practice presentation or when a patient is being monitored in hospital. The score ranges from 0 (best) to 23 (worst).
  Median time is estimated by Kaplan-Meier method, with dead patients being censored at the maximum follow-up time in the study.
Time Frame: 29 days
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 286 | 145
days | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 5.0]
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Test type: Superiority; p = 0.869, Proportional hazards model; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.84 to 1.23] — Between group comparison using competing risk framework. A hazard ratio > 1 favors the ruxolitinib 5 mg arm

12. Secondary Outcome: Change From Baseline in NEWS2 Score
Description: The National Early Warning Score 2 (NEWS2) is based on a simple aggregate scoring system in which a score is allocated to physiological measurements, already recorded in routine practice presentation or when a patient is being monitored in hospital. The score ranges from 0 (best) to 23 (worst). At each visit, only patients with a value at both baseline and the respective visit are included.
  A negative change from baseline in NEWS2 score is a favorable outcome.
Time Frame: Baseline, Days 3, 5, 8, 11, 15, and 29
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
score on scale
  Day 3: number analyzed (Participants) | 264 | 135
  Day 3 | -0.7 (1.91) | -0.6 (2.13)
  Day 5: number analyzed (Participants) | 230 | 120
  Day 5 | -1.0 (2.02) | -0.8 (2.19)
  Day 8: number analyzed (Participants) | 175 | 91
  Day 8 | -1.3 (2.25) | -1.3 (2.60)
  Day 11: number analyzed (Participants) | 113 | 66
  Day 11 | -1.1 (2.70) | -1.3 (2.74)
  Day 15: number analyzed (Participants) | 257 | 132
  Day 15 | -1.9 (2.34) | -2.2 (2.35)
  Day 29: number analyzed (Participants) | 234 | 122
  Day 29 | -2.3 (2.37) | -2.5 (2.17)

13. Secondary Outcome: Change From Baseline in SpO2/FiO2 Ratio
Description: Change from baseline in peripheral oxygen saturation / fraction of inspired oxygen ratio (SpO2/FiO2 ratio). At each visit, only patients with a value at both baseline and the respective visit are included.
  A positive change from baseline in SpO2/FiO2 ratio is a favorable outcome.
Time Frame: Baseline, Day 15, Day 29
Population: Randomized participants with a valid assessment of the outcome measure.
Measure: Mean (Standard Deviation); unit: no units
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
no units
  Day 15: number analyzed (Participants) | 260 | 132
  Day 15 | 90.110 (104.4783) | 106.766 (100.9778)
  Day 29: number analyzed (Participants) | 232 | 124
  Day 29 | 105.553 (98.2452) | 109.710 (95.4279)

14. Secondary Outcome: Proportion of Patients With no Oxygen Therapy
Description: Proportion of patients with no oxygen therapy (defined as oxygen saturation ≥ 94% on room air) at Days 15 and 29. Analyses are cumulative, thus analysis on each day includes all events till that day.
  Patients with missing data at Day 15 and/or Day 29 are excluded from the analysis.
Time Frame: Day 15, Day 29
Population: Randomized participants with a valid assessment of the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
Participants
  Day 15: number analyzed (Participants) | 274 | 140
  Day 15 | 255 | 133
  Day 29: number analyzed (Participants) | 269 | 139
  Day 29 | 262 | 136
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg vs Placebo; Day 15; Test type: Superiority; p = 0.325, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.23 to 1.63] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Placebo; Day 29; Test type: Superiority; Regression, Logistic — P-value was not estimable because >97% patients fall into one category (responders) in both groups, and very few patients fall into the other one (non-responders), which made the logistic regression model fail to converge even with Firth's correction; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.25 to 5.40] — Comparison is ruxolitinib 5 mg/placebo. An odds ratio > 1 favors the ruxolitinib 5 mg arm

15. Post Hoc Outcome: All Collected Deaths
Description: Deaths in the safety population were evaluated in all participants who received at least one dose of double-blind treatment.
  Total deaths were evaluated in all participants randomized.
Time Frame: 29 days
Population: Clinical database population - all randomized participants
Measure: Number; unit: participants
Arm/Group | Ruxolitinib 5 mg | Placebo
Number analyzed (Participants) | 287 | 145
participants
  Deaths in the safety population: number analyzed (Participants) | 281 | 143
  Deaths in the safety population | 9 | 3
  Total deaths | 9 | 3

ADVERSE EVENTS:
Time Frame: From first dose of double-blind treatment and up to the last study visit (Day 29).
Description: Adverse events are considered as treatment-emergent if the event started after the first dose of double-blind treatment or the event was present prior to start of double-blind treatment but increased in severity based on preferred term and up to the last study visit (Day 29).
  Adverse events and all-cause mortality are evaluated in the Safety Set that includes all participants who received at least one dose of double-blind treatment.
Arm/Group | Ruxolitinib 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 9/281 | 3/143
Serious Adverse Events (participants affected / at risk) | 31/281 | 15/143
Other Adverse Events (participants affected / at risk) | 113/281 | 62/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 5 mg (N=281) | Placebo (N=143)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Adverse event (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Performance status decreased (General disorders) | 1 | 0
Antibiotic associated colitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 8 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 5 mg (N=281) | Placebo (N=143)
Leukocytosis (Blood and lymphatic system disorders) | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 6 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 21 | 12
Nausea (Gastrointestinal disorders) | 6 | 11
Asthenia (General disorders) | 6 | 0
Fatigue (General disorders) | 10 | 2
Pyrexia (General disorders) | 6 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Alanine aminotransferase increased (Investigations) | 17 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 3
Transaminases increased (Investigations) | 7 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 | 3
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 23 | 11
Anxiety (Psychiatric disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypertension (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT04362137/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04362137/SAP_001.pdf